CLINICAL TRIAL: NCT02225626
Title: Effect of Food on the Pharmacokinetics of BI 1060469 (Formulation Tablet) in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1333.44; 2014-001960-37 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-08-25; First posted 2014-08-26 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Healthy

ARMS (2):
- BI 1060469 fed (Experimental): tablet, oral administration with 240 mL water 30 minutes after subject is served a standardised high-caloric high-fat administr
  Interventions: Drug: BI 1060469; Drug: Other: standard breakfast
- BI 1060469 fasted (Experimental): tablet, oral administration with 240 mL of water after an overnight fast of at least 10 h
  Interventions: Drug: BI 1060469

INTERVENTIONS:
Drug: BI 1060469 — tablet, oral administration with 240 mL of water after an overnight fast of at least 10 h
  Arms: BI 1060469 fasted
Drug: BI 1060469 — tablet, oral administration with 240 mL water 30 minutes after subject is served a standardised high-caloric high-fat administration
  Arms: BI 1060469 fed
Drug: Other: standard breakfast — tablet, oral administration with 240 mL water 30 minutes after subject is served a standardised high-caloric high-fat administration
  Arms: BI 1060469 fed

SUMMARY:
Effect of food on the pharmacokinetics of BI 1060469 (formulation tablet) in healthy male subjects as well as to investigate pharmacokinetics, safety and tolerability

ELIGIBILITY:
Inclusion criteria:

* healthy male according to the investigator´s assessment, based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead ECG, and clinical laboratory tests
* Age of 18 to 50 years (incl.)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation

Exclusion criteria:

* Any finding in the medical examination (including blood pressure (BP), pulse rate (PR) or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure greater than 140 mmHg or diastolic blood pressure greater than 90 mmHg
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Repeated measurement of pulse rate < 50 bpm and > 90 bpm at screening
* Serum creatinine laboratory value outside the normal range
* estimated glomerular filtration rate (eGFR) according to CKD-EPI-Creatinine Formula < 90 ml/ min
* Current or history of relevant kidney, urinary tract diseases or abnormalities (i.e. nephrolithiasis, hydronephrosis, acute or chronic nephritis, renal injury, renal failure, infections)
* Any evidence of a concomitant disease judged as clinically relevant by the investigator Repeated measurement of pulse rate < 50 bpm and > 90 bpm at screening
* Serum creatinine laboratory value outside the normal range
* estimated glomerular filtration rate (eGFR) according to CKD-EPI-Creatinine Formula < 90 ml/ min
* Current or history of relevant kidney, urinary tract diseases or abnormalities (i.e. nephrolithiasis, hydronephrosis, acute or chronic nephritis, renal injury, renal failure, infections)
* Any evidence of a concomitant disease judged as clinically relevant by the investigator

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
AUC 0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | up to 6 days after last drug administration
Cmax (maximum measured concentration of the analyte in plasma) | up to 6 days after last drug administration
Frequency of subjects with drug-related adverse events | up to 7 days after last drug administration

SECONDARY OUTCOMES:
AUC0-infinity (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 6 days after last drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1333.44.1 Boehringer Ingelheim Investigational Site, Ingelheim, Germany